CLINICAL TRIAL: NCT05877651
Title: A Single-center, Phase I Clinical Study to Evaluate the Safety and Tolerability of Multi-Antigen Stimulated Cell Therapy-I Injection (MASCT-I) in Patients With Metastatic or Recurrent Solid Tumors Who Failed Standard Therapy.
Brief Title: MASCT-I in Patients With Metastatic or Recurrent Solid Tumors Who Failed Standard Therapy.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HRYZ Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MASCT-I-2001
Record Dates: First submitted 2023-05-09; First posted 2023-05-26 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MASCT-I injection (Experimental): MASCT-I injection
  Interventions: Biological: MASCT-I injection

INTERVENTIONS:
Biological: MASCT-I injection — The final products of MASCT-I technology are dendritic cells (DC) and effector T cells

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of MASCT-I in patients with metastatic or recurrent solid tumors who failed standard therapy.

DETAILED DESCRIPTION:
The study is divided into two stages. The first stage is divided into two groups, both of which adopted 3+3 design. The first group is given MASCT-I by administration method 1, and the second group is given by method 2. One of the administration method will be used in the second stage according to DLT and adverse events found in the first stage.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years and ≤70 years.
* 2. Written informed consent was obtained.
* 3. Pathologically confirmed solid tumors (including but not limited to soft tissue sarcoma/osteosarcoma, urothelial carcinoma, colorectal cancer), metastatic or recurrent, and failed or intolerant to standard therapy, or lack of effective treatment; Urothelial carcinoma including renal pelvic carcinoma, bladder cancer, ureteral carcinoma or urethral carcinoma.
* 4. ECOG performance status of 0-1.
* 5. Estimated life expectancy ≥ 6 months.
* 6. Patients must have at least one measurable lesion defined by RECIST 1.1.
* 7. At least 4 weeks after the end of the last anti-tumor treatment before the 1st apheresis;
* 8. Patients with organ function as defined below (any blood components and growth factors are not allowed within 14 days before apheresis) :

  1. Leukocytes ≥ 3.0 x 10^9/L;
  2. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L;
  3. Platelets ≥ 100 x 10^9/L;
  4. Hemoglobin ≥ 90g/L;
  5. Serum albumin ≥ 3.0g/dL;
  6. Total bilirubin≤1.5×ULN; ALT/AST≤1.5×ULN (patients with liver metastasis or liver cancer, ≤5×ULN);
  7. Creatinine clearance ≥50mL/min (Cockcroft -Gault formula);
  8. Serum urea nitrogen/urea and creatinine ≤1.5×ULN (patients with urothelium carcinoma, ≤2.5×ULN);
* 9. Patients with potential fertility need to use a medically approved contraceptive measure (such as intrauterine device, contraceptive pill or condom) during the study treatment period and within 3 months after the end of the study treatment period; The serum or urine HCG test must be negative within 7 days before the study was included; And must be non lactating.

Exclusion Criteria:

* 1. Organ transplanters;
* 2. Allergic to sodium citrate or human albumin;
* 3. Patients who have undergone major surgery within 30 days before 1st apheresis (according to the investigator's definition);
* 4. Patients with uncontrolled cardiac symptoms or diseases, such as: (1) heart failure of NYHA class 2 or higher (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
* 5. Patients have received radiotherapy, hormonotherapy, surgery or targeted therapy, or immunotherapy, and less than 4 weeks before the 1st apheresis;
* 6. Patients have active infection or fever of unknown cause during screening and before 1st apheresis is more than 38.5 degrees (patients with fever caused by cancer is eligible for enrollment according to investigator's judgement);
* 7. Patients have clinically symptomatic central nervous system metastases (e.g., brain edema, need for hormonal intervention, or progression of brain metastases). Patients have previously received treatment for brain or leptomeningeal metastases were eligible if they have been clinically stable for at least 2 months and stopped systemic hormone therapy (dose >10mg/day prednisone or other therapeutic hormones) for more than 2 weeks;
* 8. Patients were using immunosuppressive agents or systemic or absorbable local hormones to achieve immunosuppressive purposes (dose > 10mg/day prednisone or other therapeutic hormones) and were still using them within 2 weeks before enrollment.
* 9. Systematic or long-term use of immunomodulators such as interferon, thymosin and immunosuppressive drugs such as adrenocorticosteroids in half a year; Systematic or long-term use of immunomodulators for more than three months and immunosuppressive drugs for more than one month;
* 10. Patients have received MASCT or other cellular immunotherapy in the past 1 year;
* 11. Patients have any active autoimmune disease or history of autoimmune disease;
* 12. Patients with other malignant tumors (except cured skin basal cell carcinoma, thyroid carcinoma and cervical carcinoma in situ) within 5 years before enrollment or at enrollment;
* 13. Patients with active tuberculosis;
* 14. Known active hepatitis B virus (except for liver cancer) or hepatitis C virus infection, and/or HIV or syphilis infection;
* 15. Patients are receiving other systemic antineoplastic therapy or currently enrolled in other clinical study, or have participated in an investigational drug trial or used an investigational device within 4 weeks before 1st apheresis, or have not recovered from toxicity of the last treatment (adverse events should be grade 1 or less according to CTCAE criteria or return to the baseline before treatment);
* 16. According to investigator's judgement, those who are not suitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Adverse events and serious adverse events related to MASCT-I | 8 weeks
  Assessed by CTCAE V5.0

SECONDARY OUTCOMES:
Adverse events and serious adverse events related to MASCT-I | 2 years
  All adverse events and serious adverse events related to MASCT-I during the study
Immune response to tumor-associated antigens | 2 years
  Measured by enzyme linked immunospot assay
Concentration of Cytokines (IFNγ、IL2、IL4、IL6、IL10 and TNF) | 2 years
  Measured by flow cytometry or other methods

OTHER OUTCOMES:
Progression-Free Survival (PFS) | 2 years
  The length of time from enrollment until the time of progression of disease
Objective Response Rate (ORR) | 2 years
  Percentage of patients with PR and CR in the total number of patients.
Disease Control Rate (DCR) | 2 years
  Disease control rate is defined as the number of patients with a best overall response of complete response (CR), partial response (PR), or stable disease (SD) based on RESIST v1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China